CLINICAL TRIAL: NCT06281808
Title: Image Quality and Diagnostic Accuracy of Photon Counting Computed Tomography of the Upper and Lower Extremity
Brief Title: Photon Counting Detector CT Image Quality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reto Sutter, MD (Other)
Responsible Party: Sponsor-Investigator, Reto Sutter, MD, Prof. Dr. med. Reto Sutter, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R490
Record Dates: First submitted 2024-02-05; First posted 2024-02-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Diagnostic Imaging; Tomography, X Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Photon Counting Detector CT (Experimental): PCD CT
  Interventions: Device: Photon Counting Detector CT

INTERVENTIONS:
Device: Photon Counting Detector CT — Photon counting detector CT scan with dose arbitrarily reduced compared to EID CT scan (e.g., half the dose of EID CT)

SUMMARY:
This study aims to compare subjective image quality and diagnostic accuracy of a photon counting detector computed tomography (PCD-CT) scanner compared with an energy integrating detector (EID)-CT scanner as the reference standard.

DETAILED DESCRIPTION:
Computed tomography (CT) imaging plays a key role in diagnostic radiology, and is particularly valuable in assessing a myriad of musculoskeletal conditions (e.g. trauma, degenerative disorders, post-surgical follow-up, inflammatory diseases).

The vast majority of today's CT scanners are equipped with an energy-integrating detector (EID), which converts energy of incoming X-ray photons in a two-step process into electric signals: First, scintillators generate visible light, which in turn is converted to the electric signal by photodiodes.

Recently, photon-counting detector computed tomography (PCD-CT) scanners became commercially available and have been introduced to improve imaging performance through direct transformation of X-ray photons into electron hole pairs upon absorption in a semiconductor layer, generating an electrical signal proportional to the photon energy.

Current literature has shown that PCD-CT can offer higher spatial resolution, increased contrast-to-noise ratio, higher dose-efficiency, and inherent multi-spectral imaging capacity.

Moreover, the results from cadaver studies suggest that PCD-CT can preserve image quality with reduced radiation dose.

However, data on the diagnostic accuracy of PCD-CT compared to EID-CT is currently limited in the field of musculoskeletal radiology.

In addition to conventional CT acquisition, multi-spectral CT imaging in patients with gout and after trauma, is used in clinical routine to delineate materials with a specific absorption coefficient: in gout, urate crystals can be visualized, while after trauma, bone marrow edema can be detected. For EID-CT, different techniques for multi-spectral CT imaging are available (e.g. fast kV switching, dual source CT) which are widely used in clinical routine. Multi-spectral imaging is also inherently available for recently introduced PCD-CT. However, data on diagnostic accuracy of multi-spectral PCD-CT is currently lacking.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted for non-contrast enhanced CT scan of the upper or lower extremity at the radiology department of Balgrist University Hospital
* Signed general consent ("Information zur Weiterverwendung gesundheitsbezogener Daten und Proben zu Forschungszwecken")
* >18 years of age
* Written consent to participate in this study

Exclusion Criteria:

* Clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Women: pregnancy
* Age below 18 years
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to consent and/or follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc. of the subject
* Enrolment of the PI, his/her family members, employees and other dependent persons
* Body mass above 200 kg.
* Body mass below 31 kg.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-28 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Image Quality PCD CT | 2 years
  Likert scale based - 5 point Likert scale (0 = worst, 5 = best)
  Visual gradings of PCD-CT image quality. Image quality will be assessed by teams of experienced musculoskeletal radiologists. Images from consistent sets of intra-subject PCD-CT and EID-CT data will be presented to derive the primary outcome data, in particular using visual analog scales (Likert-Scales). Inter-reader reliability will be assessed.
Diagnostic Accuracy PCD CT | 2 years
  This will involve the calculation of sensitivity, specificity, positive predictive value, negative predictive value, and overall accuracy. The EID-CT image interpretation of the attending radiologists, as documented in the written report, will serve as reference standard against which the performance of PCD-CT will be compared. In cases with inconclusive written reports and image findings of EID-CT, a review committee consisting of experienced radiologists (e.g., other attending radiologists, chief of radiology) will be convened, and consensus reading including clinical correlation by consulting with the treating physicians and specialists involved in the patient's care will be done. Diagnostic confidence will be additionally analyzed for PCD-CT scans on a Likert-Scale. Inter-reader reliability will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No